CLINICAL TRIAL: NCT06813326
Title: Interest of Nurse Participation During Epicutaneous-cavity Catheter Placement in Neonatal Intensive Care
Acronym: IPICAVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AOI 2023 SATURNIN
Record Dates: First submitted 2025-01-14; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Premature Birth
Keywords: newborn; neonatal intensive care; percutaneous central venous catheter; nurse; pain; shots
MeSH Terms: conditions — Premature Birth; Pain | interventions — Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4 hand (Experimental): At D1, on the first attempt, the KTEC will be inserted by an I(P)DE/physician pair served by the nurse in charge of the child (whatever their level of experience) using the standard method, with no limit to the number of injections.
  At D2, if KTEC insertion fails at D1, a second attempt will be made, respecting the newborn's randomization arm. This second attempt must be carried out by an I(P)DE/doctor pair, with the nurse having a minimum of three years' seniority in a neonatal intensive care unit, and whose expertise will ensure successful insertion, with the number of injections limited to five.
  At D3, in the event of a further failure at D2, a third and final attempt will be made by a senior doctor, with no limit on the number of injections (to encourage success), in line with current department practice.
  Translated with DeepL.com (free version)
  Interventions: Procedure: catheter insertion
- 2 hand (Active Comparator): At D1, on the first attempt, the KTEC will be inserted by the doctor alone (junior or senior, depending on availability), assisted by the nurse responsible for the child, using the standard method, with no limit on the number of injections.
  On D2, if KTEC insertion fails on D1, a second attempt will be made, respecting the newborn's randomization arm. This second attempt must be made by a senior doctor in the department, whose expertise will help ensure successful insertion, with the number of injections limited to five.
  At D3, in the event of a further failure at D2, a third and final attempt will be made by another senior doctor, with no limit on the number of injections (to encourage success), in line with the department's current practice.
  Translated with DeepL.com (free version)
  Interventions: Procedure: catheter insertion

INTERVENTIONS:
Procedure: catheter insertion — success of catheter insertion

SUMMARY:
To meet the needs of newborns in neonatal intensive care and ensure long-term venous access, a percutaneous central venous catheter (KTEC) is inserted. According to the recommendations of the French Society of Hospital Hygiene, the placement of this device is the responsibility of a medical professional. It may require several attempts to ensure the success of the procedure.

The pain associated with the needle insertion is generally controlled, but with repeated attempts, the newborn may become agitated, cry, and be difficult to calm. The study by Courtois et al. showed that pain in infants under 45 weeks of gestational age increased with the number of attempts. Acute and repeated pain in newborns can lead to trauma and disturbances in psychological, cognitive, and motor development.

In the neonatal intensive care unit (NICU) at the University Hospital of Clermont-Ferrand, the procedure is performed by the physician alone (i.e., "two hands"), whereas in other NICUs in France, the procedure is systematically performed by a nurse/physician team (i.e., "four hands"). However, no comparative study has been conducted to date to assess the impact of this "four hands" approach on the number of needle attempts and the pain experienced by the newborn.

The investogator hypothesize that the training and participation of the nurse (pediatric nurse) during the placement of the KTEC, in collaboration with the physician, could reduce the number of needle attempts and the newborn's pain. Therefore, the investigator aim to conduct a randomized, monocentric pilot study in the neonatal intensive care unit at the University Hospital of Clermont-Ferrand.

DETAILED DESCRIPTION:
In the neonatal intensive care unit (NICU) of the University Hospital of Clermont-Ferrand (63), the study will begin with the training of a group of nurse practitioners (I(P)DE) to perform KTEC insertions in pairs over a six-month period. After this training, if a KTEC insertion is required, the investigator will ask the parents or guardians of eligible newborns for their consent to participate in the IPICAVE study (pre-inclusion visit).

If they agree, inclusion/randomization will take place after the parents or legal guardians sign the informed consent form for study participation.

The inclusion period will last for 18 months, and the study participation for each newborn will begin with the first needle insertion during the procedure and end at the conclusion of the dressing change after successful KTEC insertion or upon the last needle insertion if the attempt fails. During the KTEC insertion, the responsible I(P)DE will complete a data collection form to assess the various study criteria.

ELIGIBILITY:
Inclusion Criteria:

* Newborns born between 25 and 42 weeks of amenorrhea requiring KTEC insertion
* Newborn whose parents or guardians have been informed of the study and are capable of providing informed consent to participate in the research.
* Informed consent obtained from parents or guardians
* Parents of legal age (≥18 years)

Exclusion Criteria:

* Parents under guardianship or curatorship, deprived of liberty or under court protection
* Parents who do not speak or understand French
* Newborn born under X

Max Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-02-04 (Estimated); Study Completion 2027-02-04 (Estimated)

PRIMARY OUTCOMES:
Successfull of KTEC insertion | within day 3
  Total number of injections until successful KTEC insertion.

SECONDARY OUTCOMES:
success rate of the procedure. | within day 3
  Success or failure of KTEC insertion.

OTHER OUTCOMES:
pain evaluation | within day 3
  Average and maximum pain during injections, measured by hetero-evaluation scales
number of insertion attempts in cases of previous failure | within day 3
  Total number of previous unsuccessful placement attempts
procedure time | within day 3
  procedure time in minutes
Study the factors associated with the total number of bites | within day 3
  number of bites according to the occurrence or non-occurrence of state of consciousness (awake or sedated newborn)
Study factors associated with average and maximum pain in newborns | within day 3
  average and maximum pain according to state of gestational age (in weeks of amenorrhea: ˂29 , 29 to 32, 33 to 36, 37 to 42, and >42)
hemoglobin levels | within day 3
  Percentage change in hemoglobin between two consecutive days (dependent variable) and number of injections performed between the two hemoglobin measurements (independent variable)
Study the factors associated with the total number of bites | within day 3
  number of bites according to catheter type (Premicath, Epicutaneocave, Nutriline twinflow)
Study factors associated with average and maximum pain in newborns | within day 3
  average and maximum pain according to insertion site (left/right upper limb, left/right lower limb, skull)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie SATURNIN LENOBLE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No